CLINICAL TRIAL: NCT01553617
Title: Efficacy and Safety of Perioperative Infusion of 6 % Hydroxyethyl Starch 130/0.4 in an Isotonic Electrolyte Solution (VolulyteTM) vs. 5% HSA as Volume Replacement Therapy During Cardiac Surgery for Adult Patients
Brief Title: VolulyteTM in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VOLU-010-C P4
Record Dates: First submitted 2012-03-07; First posted 2012-03-14 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volulyte (Experimental): 6 % hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution (VolulyteTM)
  Interventions: Drug: 6% hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution (VolulyteTM)
- Human serum albumin (Active Comparator): Human serum albumin (HSA 50g/L)
  Interventions: Drug: Human serum albumin

INTERVENTIONS:
Drug: 6% hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution (VolulyteTM) — Study drug will be given as part of priming of the ECC and for volume therapy up to the maximum dosage of 50 mL/kg body weight/day
  Arms: Volulyte
Drug: Human serum albumin — Control drug will be given as part of priming of the ECC and for volume therapy up to the maximum dosage of 50 mL/kg body weight/day
  Arms: Human serum albumin

SUMMARY:
The study will compare the efficacy and safety of VolulyteTM and human albumin in elective open-heart surgery in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female adult patients
* undergoing primary elective cardiac surgery applying extracorporeal circulation
* signed written informed consent

Exclusion Criteria:

* known contraindication against scheduled medication
* pre-operative acute normovolaemic haemodilution or preoperative autologous blood donation
* planned systemic hypothermia (body temperature < 30°C)
* expected time on ECC ≥ 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Calculated red blood cell loss | up to 3rd postoperative day

SECONDARY OUTCOMES:
Haemodynamics | up to 3rd postoperative day
Fluid input/output | up to 3rd postoperative day
  Quantity of total fluids administered and excreted or lost from beginning of anaesthesia until 3rd postoperative day
Use of vasoactive and inotropic drugs | up to 3rd postoperative day
  Type and amount of vasoactive and inotropic drugs administered from beginning of anaesthesia until 3rd postoperative day
Laboratory parameters | up to day 28 after surgery
  Serum creatinine concentration at day 28 after surgery
Laboratory parameters | up to 3rd postoperative day
  set of standard laboratoy parameters before surgery and postoperatively until 3rd postop day

CONTACTS AND LOCATIONS:
Overall Officials: David C Mazer, Principal Investigator — St. Michael's Hospital, Department of Anaesthesia, 30 Bond Street, Toronto, Ontario, M5B 1W8, Canada
Locations (5):
- Canada (5):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario